CLINICAL TRIAL: NCT02426242
Title: Observational Evaluation of Risk Factors Regarding Extubation Failure in Severe Brain-injured Patients
Brief Title: Evaluation of Risk Factors Regarding Extubation Failure in Severe Brain Injured Patients.
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC13_0354
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2015-04

CONDITIONS: Severe Brain Injury
Keywords: brain-injury; extubation
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICU PATIENTS: Patients with brain-injury
  Interventions: Other: Collection of medical data from ICU patients

INTERVENTIONS:
Other: Collection of medical data from ICU patients — A code will be applied to each patient included. Medical data such as demography, ISS, clinical exam at time of extubation, extubation failure, tracheotomy, will be collected during ICU stay.

SUMMARY:
Severe brain-injured patients require prolonged mechanical ventilation. Weaning these patients from mechanical ventilation is challenging. During neurologic recovery, brain injured patients usually present satisfactory respiratory autonomy. However, the exact timing of extubation is unknown and is frequently delayed because of potential inhalation.

To date, there are no clinical signs available in the current literature that can help the attending physician in the decision-making process of extubation in brain-injured-patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with brain-injury (traumatic brain injury, subarachnoid haemorrhage, stroke, intracerebral hemorrhage, brain tumour) requiring ≥ 48 hours of mechanical ventilation after admission

Exclusion Criteria:

* Pregnant women
* Patient consent withdrawal

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized in ICU for severe brain injury
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Extubation failure | In the 48 hours following extubation
  Extubation failure is regarded as the need of intubation in the 48 hours following extubation Establish clinial signs before extubation that can predict extubation failure Realization of a systematic clinical examination by the attending physician before performing extubation in severe brain-injured patients

SECONDARY OUTCOMES:
Impact of extubation failure | Median 14 days after Intensive Care Unit (ICU) admission
  Impact of extubation failure on
  * Duration of mechanical ventilation
  * Length of ICU stay
  * Mortality Describing reasons

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël Cinotti, MD, Principal Investigator — Nantes University Hospital
Locations (3):
- France (3):
  - Angers University Hospital, Angers
  - Nantes University Hospital, Nantes
  - Rennes University Hospital, Rennes